CLINICAL TRIAL: NCT03927183
Title: Extended Support Within a Person-centred Practice After Surgery: a Quasi- Experimental Study for Persons With Pituitary Tumours
Brief Title: Extended Support for Persons With Pituitary Tumours After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GoPT
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Pituitary Tumor Benign; Surgery
Keywords: Person-centred care; Clinical pathway; Intervention; Quasi-experimental

STUDY DESIGN:
Intervention Model Description: A quasi- experimental study with non-equivalent control group design, pretest-posttest study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Person-centred practice (Other): Person-centred care
  Interventions: Other: person-centred practice

INTERVENTIONS:
Other: person-centred practice — The structure and content of the intervention is constructed on principles for person-centredness. Each patients in the intervention are allocated a hospital-initiated nurse care manager during one year after surgery. Self-management support is primarily conducted between the patient and the nurse care manager. The primary goal of the support is to facilitate patients own resources in managing illness and health education on e.g. physical activity and diet. The support also comprises patient-held documentation and health plan. Other components of the intervention comprise accessibility and continuity which is secured by a structured clinical care pathway with planned care and defined care contacts. The patient has continuous access to the nurse care manager by telephone and face-to-face contact according to a structured follow-up plan. An interdisciplinary team as well as a patient education program constitutes distinct parts of the support during the year after surgery.

SUMMARY:
Patients with pituitary tumours often live with life-long consequences of their disease. Treatment options include surgery, radiotherapy and medical therapy. Symptoms associated with the tumour and/or its treatment affects several areas of life. The year after pituitary surgery constitutes an important time-period with medical evaluations of surgery and decisions on hormonal substitution. The development and evaluation of extended patient support during this time-point is limited. Care based on person-centredness has exclusively been promoted which comprises a care where care providers inquire how patients view their health situation and what their needs, resources, and preferences are. Person-centredness focuses on preserving patient autonomy, function, and well-being and strives to emphasize patient involvement through equalizing power between health care professionals and the patient with the main goal of an enhanced health situation. The aim of the study is to evaluate if a support within a person-centered care practice one year after surgery increases wellbeing for patients with pituitary tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Pituitary tumour; adenoma or craniopharyngioma
2. Planned neurosurgery due to pituitary tumour

Exclusion Criteria:

1. Pituitary carcinomas
2. Health conditions which may restrain the understanding of the study and/or the ability to adhere to the protocol for example decreased cognitive functions or drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Self- perceived psychological wellbeing | From date of inclusion until the date of one year follow up after surgery
  The outcome is assessed with The Psychological General Well-being scale (PGWB), a questionnaire with 22 items, comprising six subscales: anxiety, depression, positive well-being, self-control, general health and vitality. The Swedish version of the questionnaire is valid. Total score of 132 is an overall score of the values from each item (score 1-6 for each item). Higher value is indicative for better psychological well-being. A sum score for each subscale can be calculated, minimum and maximum score; anxiety (5-30), depression (3-18), positive well-being (4-24), self-control (3-18), general health (3-18) and vitality (4-24).

SECONDARY OUTCOMES:
Person-centred content in medical records | From date of inclusion until the date of one year follow up after surgery
  Degree of person-centredness in medical records according to dimensions in a protocol to review content in medical records.
Self-reported health assessed with EQ-5D-5L | From date of inclusion until the date of one year follow up after surgery.
  Self-reported health is measured with the EuroQual-5Dimensions-5Levels questionnaire (EQ- 5D- 5L). The questionnaire comprises 1 item per dimension. The dimensions of importance for health which are included are; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients rate each item on a scale ranging from 1 (no problems) to 5 (extreme problems/unable to). A unique health state is defined by combining 1 level from each of the 5 dimensions. The questionnaire also includes EQ-VAS, in which the patients grade their current health status on an analogue scale from 0 (worst health) to 100 (best health).
Fatigue assessed with the Multidimensional Fatigue Inventory (MFI-20) | From date of inclusion until the date of one year follow up after surgery.
  Within MFI-20 general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue comprises five dimensions of fatigue. Fatigue in the preceding seven days is rated on a 5-point Likert scale from "yes, that is accurate to "no, that is not accurate". Subscale scores range from 4-20, where a high score represents greater fatigue.
Quality of care assessed with the Quality from the Patient Perspective questionnaire | From date of inclusion until the date of one year follow up after surgery
  The outcome is assessed with the questionnaire Quality from the Patient Perspective. The questionnaire comprises four dimension Identity-oriented approach (13 items) and the sociocultural atmosphere (5 items), medical- technical competence (4 items) and physical-technical condition (3 items). Two kinds of assessments are being made at each item: whether things were being done (perceived reality) and whether the right things were being done (subjective significance). Items are rated on a four-point response scale ranging from 1 (do not agree at all) to 4 (completely agree). Each item also has a response option of "not applicable". Subscales can be reported item by item or combined in a subscale score (average of all responses within the subscale).
Level of general self-efficacy assessed with the General Self-Efficacy scale | From date of inclusion until the date of one year follow up after surgery
  General self-efficacy measures confidence in one's ability to handle difficult challenges in life. It includes 10 items, which are rated on a four- point Likert scale giving a summary score of 40 for the total scale (10-40).

OTHER OUTCOMES:
Clinical observations of pulse rate | From date of admission to inpatient care after surgery until the date of discharge, up to 60 days of hospitalization
  Frequency of documented pulse rate during hospitalization. The medical records are reviewed retrospectively.
Quality of care assessed as documented information in medical records on current medication at a daily basis and at discharge: rating | From date of admission to inpatient care after surgery until the date of discharge, up to 60 days of hospitalization
  All information in the medical records during hospitalization are reviewed retrospectively. Rating is made regarding the presence (yes or no) of information on current medication at a daily basis and at discharge.
Quality of care assessed as documented information in medical records on planned medical care at discharge: rating | From date of admission to inpatient care after surgery until the date of discharge, up to 60 days of hospitalization
  All information in the medical records during hospitalization are reviewed retrospectively. Rating is made regarding the presence (yes or no) of information on planned medical care at discharge.
Clinical observations of weight | From date of admission to inpatient care after surgery until the date of discharge, up to 60 days of hospitalization
  Frequency of documented clinical observations of weight (kg) during hospitalization. The medical records are reviewed retrospectively.
Clinical observations of respiratory rate | From date of admission to inpatient care after surgery until the date of discharge, up to 60 days of hospitalization
  Frequency of documented clinical observations of respiratory rate during hospitalization. The medical records are reviewed retrospectively.
Clinical observations of body temperature | From date of admission to inpatient care after surgery until the date of discharge, up to 60 days of hospitalization
  Frequency of documented clinical observations of body temperature (degrees celsius) during hospitalization. The medical records are reviewed retrospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Jakobsson Ung, professor, Principal Investigator — Göteborg University
Locations (1):
- Department of Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No